CLINICAL TRIAL: NCT01275183
Title: A Pilot Study of Raltegravir and Cisplatin in Squamous Cell Carcinoma of the Head and Neck
Brief Title: Pilot Study of Raltegravir and Cisplatin in Squamous Cell Carcinoma of Head and Neck
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1012; NCI-2012-00914 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-01-06; First posted 2011-01-12 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; SCC; head and neck; squamous cell; nasopharyngeal
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Raltegravir Potassium; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir and cisplatin (Experimental)
  Interventions: Drug: raltegravir and cisplatin

INTERVENTIONS:
Drug: raltegravir and cisplatin — Cisplatin, intravenous, 30 mg/m2, days 2 and 16, 1 to 2 hours
  Raltegravir, oral,400 mg, twice per day, days 1 through 5 or days 15 to 19
  Part 2 (optional): Docetaxel, intravenous, 75 mg/M2, day 2, every 21 days, 3 to 6 cycles
  Part 2 (optional): Cisplatin, intravenous, 75 mg/M2, day 2, every 21 days, 3 to 6 cycles
  Part 2: (optional): Raltegavir, oral, 400 mg, twice per day, days 1 through 5, 3 to 6 cycles
  Other Names: MK-0518; Isentress; raltegravir; cisplatin; docetaxel; Taxotere

SUMMARY:
The proposed study is a first-in-human pilot of a novel anti-cancer strategy: Metnase inhibition to potentiate DNA damaging chemotherapy. The investigators will conduct serial tumor biopsies in subjects with HNSCC at three timepoints: baseline, after cisplatin, and after cisplatin-raltegravir. The investigators will investigate immunohistochemical expression changes of γH2AX, Chk2, and Annexin V, three biomarkers of DNA damage and apoptosis. The study is designed to identify an intermediate signal of the potentiation of cisplatin chemotherapy by raltegravir in HNSCC, which will justify a future phase I/II study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of squamous cell carcinoma of the head and neck. All primary sites are eligible, including keratinizing nasopharyngeal carcinoma (WHO grade 1 or 2) and carcinoma of unknown primary.
* Either the primary site or a metastatic locoregional tumor deposit (eg. lymph node, parotid gland, subcutaneous nodule) must be amenable to repeat, in-office biopsy by a head and neck surgeon.
* The patient must be considered an appropriate candidate for cisplatin chemotherapy by a medical oncologist. Acceptable indications include induction chemotherapy prior to surgery or radiation for localized disease, or palliative chemotherapy for advanced disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate bone marrow function, defined as an absolute peripheral granulocyte count of greater than 1,500 cells/mm3 and platelet count greater than 100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Adequate hepatic function with a total bilirubin less than 2 mg/dl; SGOT and SGPT less than 1.5 times the upper limit of normal; alkaline phosphatase less than 2.5 times the upper limit of normal.
* Creatinine clearance greater than or equal to 55 mL/min. Creatinine clearance will be estimated by the Cockraft-Gault formula, using actual body weight.
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment, and for at least 3 months thereafter.
* Age greater than 18.
* Able to provide written, informed consent.

Exclusion Criteria:

* No known brain metastases.
* Pregnant women or nursing mothers are not eligible for this trial.
* During the first two weekly cycles of cisplatin and raltegravir, patients may receive no other concurrent antineoplastic therapy, including chemotherapy, biologic agents or radiotherapy. For subsequent induction or palliative chemotherapy cycles, patients may receive combination cisplatin-docetaxel-raltegravir, on a three-week schedule as specified in this protocol.
* No severe medical problems, including unstable angina; myocardial infarction within the past 6 months; symptomatic congestive heart failure, NYHA grade II or higher; active infection requiring antibiotics.
* History of hypersensitivity reaction to cisplatin.
* Patient with known HIV disease.
* Any comorbid condition which would preclude full compliance with the protocol.
* Patient is less than 3 years free from another malignancy, except: a) if the other malignancy is non-melanomatous skin cancer or cervical carcinoma in situ or b) if the other primary malignancy is considered clinically insignificant and is requiring no active intervention.
* Peripheral neuropathy greater than or equal to grade 2.
* Ongoing treatment with rifampin, phenytoin, or phenobarbital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Gene expression modification | 3 weeks
  Expression changes of three selected tumor biomarkers (DNA damage and apoptosis) will be measured at baseline, after cisplatin alone, and after raltegravir-cisplatin. Tumor biomarkers include pChk2, Annexin V, and metnase.

SECONDARY OUTCOMES:
Clinical activity | 2 to 6 months
  Preliminary clinical activity of the combination of raltegravir and cisplatin-based chemotherapy in HNSCC will be measured by RECIST criteria. Patients who elect participation in Part 2 will undergo tumor response assessment in accordance with RECIST 1.1 criteria after every 3 cycles of cisplatin-docetaxel-raltegravir. Response rate after 3 cycles will be reported as applicable.
  Preliminary toxicity of the combination of raltegravir and cisplatin-based chemotherapy in HNSCC as measured by the grading system (0-4) of the NCI CTCAE v.4
  Baseline Metnase expression in HNSCC.
Clinical toxicity | 2 to 6 months
  Preliminary toxicity of the combination of raltegravir and cisplatin-based chemotherapy in HNSCC as measured by the grading system (0-4) of the NCI CTCAE v.4
Progression free survival and overall survival | 2 years
  Progression-free and overall survival duration will be measured from entry into the protocol, until death.
Metnase expression | 2 to 6 months
  From biopsy materials, quantitative score generated by Aperio Scanning. Digital photomicrographs will be scored for frequency and intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Houman Fekrazad, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: UNM Cancer Center — http://cancer.unm.edu